CLINICAL TRIAL: NCT00072475
Title: A Phase II Study of an Oral VEGF Receptor Tyrosine Kinase Inhibitor (PTK787/ZK222584) (IND #66370, NSC #719335) in Myelodysplastic Syndrome (MDS)
Brief Title: Vatalanib in Treating Patients With Primary or Secondary Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-10105; U10CA031946 (NIH); CALGB-10105; CDR0000339810 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; refractory anemia; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Anemia, Refractory | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vatalanib (Experimental): Adult patients with MDS receive treatment with vatalanib.
  Interventions: Drug: vatalanib

INTERVENTIONS:
Drug: vatalanib — Pts registered before 1/15/05 1250 mg/day PO After 1/15/05: Start w/ 750 mg/day PO; escalate q 4 wks in absence of Grade 2 or > tox (1st increase=1000mg/day; 2nd increase 1250 mg/day)
  Other Names: PTK787/ZK 222584

SUMMARY:
RATIONALE: Vatalanib may be effective in preventing the development of leukemia in patients who have myelodysplastic syndromes.

PURPOSE: This phase II trial is studying vatalanib to see how well it works in treating patients with primary or secondary myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate, in terms of hematologic improvement and complete and partial remission, in patients with primary or secondary (therapy-related) myelodysplastic syndromes treated with vatalanib.
* Determine the time to transformation to acute myeloid leukemia (at least 20% blasts) or death in patients treated with this drug.

Secondary

* Determine the safety of this drug in these patients.
* Determine the duration of response in patients treated with this drug.
* Determine the cytogenetic response rate in patients treated with this drug.
* Determine the overall and progression-free survival of patients treated with this drug.
* Determine the incidence of infections requiring antibiotics or hospitalization or bleeding requiring red blood cell transfusions in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified* according to risk group (low grade [refractory anemia with or without ringed sideroblasts, refractory anemia with excess blasts-1, refractory cytopenia with multilineage dysplasia with or without ringed sideroblasts, myelodysplastic syndromes-unclassified, or chronic myelomonocytic leukemia-1] vs high grade [refractory anemia with excess blasts-2 or chronic myelomonocytic leukemia-2]).

NOTE: *Stratification according to risk (low vs high) does not occur after 11/30/06.

Patients receive oral vatalanib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 6 additional courses after documentation of a CR.

Patients are followed periodically for up to 5 years from study entry.

PROJECTED ACCRUAL: Approximately 144 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary or secondary (therapy-related) myelodysplastic syndromes* (MDS), including the following cellular types:

  * Refractory anemia (RA)**
  * RA with excess blasts (RAEB)-1
  * RA with ringed sideroblasts**
  * Refractory cytopenia with multilineage dysplasia
  * Refractory cytopenia with multilineage dysplasia with ringed sideroblasts*
  * MDS-unclassified**
  * MDS associated with isolated del (5q)**
  * Chronic myelomonocytic leukemia (CMML)-1 NOTE: *High-risk MDS (i.e., RAEB-2 or CMML-2) is closed to accrual as of 11/30/06

NOTE: **Accompanied with at least 1 of the following laboratory values: hemoglobin less than 10 g/dL, platelet count less than 50,000/mm3, or absolute neutrophil count less than 1,000/mm3

* No prior leukemia (i.e., 20% or greater blasts)
* No prior primary or metastatic brain tumor or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* APTT no greater than 1.5 times ULN
* INR no greater than 1.5

Renal

* Creatinine no greater than 1.5 times ULN
* Urine protein negative by urinalysis

  * Protein 1+ by dipstick allowed provided total urine protein no greater than 500 mg AND creatinine clearance at least 50 mL/min by 24-hour urine collection

Cardiovascular

* No significant cardiac or vascular events within the past 6 months, including any of the following:

  * Acute myocardial infarction
  * Unstable angina
  * Uncontrolled hypertension
  * Severe peripheral vascular disease (e.g., ischemic pain at rest or nonhealing ulcers or wounds)
  * New York Heart Association class II-IV congestive heart failure
  * Cardiac arrhythmia
  * Disseminated intravascular coagulation or other coagulopathies
  * Deep vein or arterial thrombosis
* No history of congenital long QTc syndrome or elongated QTc (> 450 msec for males or 470 for females)

Pulmonary

* No pulmonary embolism within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 3 months after study participation
* No need for full anticoagulation within the past 6 months
* No significant hemorrhage (e.g., visceral, gastrointestinal, genitourinary, or gynecological) requiring red blood cell transfusion within the past month
* No known cerebral aneurysms, other cerebrovascular malformations, or CNS bleeding
* No unhealed fractures, wounds, or ulcers

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 12 months since prior autologous stem cell or allogeneic transplantation
* More than 6 months since prior antiangiogenic agents
* More than 1 month since prior interferon for MDS
* More than 1 month since prior hematopoietic growth factors for MDS
* More than 1 month since prior epoetin alfa (EPO) for MDS
* More than 1 month since prior thalidomide for MDS
* More than 1 month since prior immunotherapy for MDS
* No concurrent prophylactic growth factors or cytokines (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], EPO or EPO-derivatives, or interleukin-11)

Chemotherapy

* No prior low-dose antimetabolites for MDS (e.g., hydroxyurea, azacitidine, or low-dose cytarabine)
* More than 12 months since prior chemotherapy for another disease* NOTE: *Not MDS or leukemia

Endocrine therapy

* More than 1 month since prior corticosteroids for MDS
* More than 1 month since prior androgens for MDS

Radiotherapy

* More than 12 months since prior radiotherapy for another disease* NOTE: *Not MDS or leukemia

Surgery

* More than 1 month since prior surgery, including needle biopsy of visceral organs and recovered

  * Bone marrow biopsy allowed
* More than 2 weeks since prior placement of a subcutaneous or tunneled venous access device (e.g., PortaCath or Hickman's catheter) and adequately healed

Other

* No prior cytotoxic therapy for MDS
* More than 1 month since prior administration of any of the following medications for MDS:

  * Danazol
  * Retinoids
  * Amifostine
  * Investigational agents
* No concurrent administration of any of the following medications:

  * Warfarin
  * Heparin
  * Derivatives of heparin
  * Other anticoagulants
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2003-12; Primary Completion 2008-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Gupta, MD, Study Chair — Veterans Affairs Medical Center - Minneapolis
Locations (68):
- United States (68):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Gupta P, Miller AA, Owzar K, et al.: Pharmacokinetics of an oral VEGF receptor tyrosine kinase inhibitor (PTK787/ZK222584) in patients with myelodysplastic syndrome (MDS): Cancer and Leukemia Group B study 10105. [Abstract] J Clin Oncol 24 (Suppl 18): A-6573, 355s, 2006.
- [Result] Gupta P, Sanford BL, Yu D, et al.: A phase II study of an oral VEGF receptor tyrosine kinase inhibitor (PTK787/ZK222584) in patients with myelodysplastic syndrome (MDS): Cancer and Leukemia Group B study 10105. [Abstract] Blood 108 (11): A-2665, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 155 participants were enrolled between December 2003 and April 2008.
Pre-assignment Details: Of the 155 participants recruited, 2 participants cancelled prior to starting treatment; 7 were determined to have AML at registration and 4 had diagnosis other than MDS. Thus 142 participants were evaluable for response and 153 for adverse events.
Groups:
- Vatalanib: Adult patients with MDS receive treatment with vatalanib.
  vatalanib: Pts registered before 1/15/05 1250 mg/day PO
  After 1/15/05: Start w/ 750 mg/day PO; escalate q 4 wks in absence of Grade 2 or > tox (1st increase=1000mg/day; 2nd increase 1250 mg/day)
Period: Overall Study
Arm/Group | Vatalanib
Started | 142
Completed | 45
Not Completed | 97
Not completed — Adverse Event | 44
Not completed — Death | 3
Not completed — Withdrawal by Subject | 46
Not completed — Patient/Investigator Decision | 4

BASELINE CHARACTERISTICS:
Population: Of the 155 participants recruited, 2 participants cancelled prior to starting treatment; 7 were determined to have AML at registration and 4 had diagnosis other than MDS. Thus 142 participants were evaluable for response
Arm/Group | Vatalanib
Number analyzed (Participants) | 142
Age, Continuous [Median (Full Range); unit: years] | 71 [27 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 133
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Response was measured by International Standardized Response Criteria for MDS
  * Complete Response: Bone marrow showing < 5% myeloblasts with normal maturation of all cell lines; Hgb > 11 g/dL (untransfused), ANC ≥1.5 K/L, PLT ≥ 100 K/L, No blasts, no dysplasia
  * Partial remission: All of the CR criteria (if abnormal at baseline), except BM evaluation. Blasts decreased by ≥ 50% over baseline. Cellularity and morphology are not relevant.
  Hematologic improvement:
  * Erythroid (HI-E): For participants with baseline HGB < 11g/dL, Major: > 2g/dL increase, transfusion independence. Minor: 1-2g/dL increase, ≥ 50% decrease in transfusion requirements
  * Platelet (HI-P): For participants with baseline PLT < 100 K/L: Major: absolute increase of > 30 K/L, transfusion independence. Minor: ≥ 50% increase (net increase of >10 K/L)
  * Neutrophil (HI-N): For participants with baseline ANC < 1.5 K/L, Major: > 100% increase (net increase > 0.5 K/L). Minor: > 100% increase (absolute increase < 0.5 K/L)
Time Frame: Duration of study (up to 5 years)
Measure: Number; unit: participants
Arm/Group | Vatalanib
Number analyzed (Participants) | 142
participants
  Complete Remission | 0
  Partial Remission | 0
  HI-E Major | 3
  HI-E Minor | 1
  HI-P Major | 2
  HI-P Minor | 1
  HI-N Major | 0
  HI-N Minor | 0

2. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the time from response (complete remission, partial remission or hematologic improvement) to progression or death of any cause. Responding and alive patients were censored at the date of last follow-up. The median DOR with 95% CI was estimated using the Kaplan Meier method.
  Response was measured by International Standardized Response Criteria for MDS (described in above outcome measure).
Time Frame: 5 yrs
Population: Per the description, only patients who achieved a response were evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vatalanib
Number analyzed (Participants) | 7
months | 6 [2 to 46]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) as the interval from the on-study date until death. OS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vatalanib
Number analyzed (Participants) | 142
months | 18.9 [15.0 to 26.8]

4. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was defined as the time from registration to progression or death of any cause. Progression free and alive patients were censored at the date of last clinical assessment. The median PFS with 95% CI was estimated using the Kaplan Meier method.
  Progression is defined as
  * For patients with <5% bone marrow blasts: ≥50% increase in blasts to >5% blasts
  * For patients with 5-10% bone marrow blasts: ≥50% increase to >10% blasts
  * For patients with 10-19% bone marrow blasts: increase to ≥20% blasts
  * One or more of the following: 50% or greater decrement from maximum remission/response levels in ANC < 1.5 K/L or PLT< 100 K/L, or reduction in HGB by at least 2 g/dL or becoming transfusion dependent
  Progression after HI: Includes one or more of the following
  * Decrement of 50% or greater from maximum response levels in ANC < 1.5 K/L or PLT < 100 K/L
  * Reduction in HGB concentration by at least 2 g/dL
  * Becoming transfusion dependent
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vatalanib
Number analyzed (Participants) | 142
months | 10.2 [7.4 to 14.74]

5. Primary Outcome: Time to Transformation to AML
Description: Time to transformation to AML is defined as the time from registration to the transformation of MDS to AML or death of any cause. Participants not meeting these criteria were censored at the date of last follow-up. This outcome was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vatalanib
Number analyzed (Participants) | 142
months | 17.2 [10.8 to 23.9]

ADVERSE EVENTS:
Groups:
- Vatalanib: After 1/15/05: Start w/ 750 mg/day PO; escalate q 4 wks in absence of Grade 2 or > tox (1st increase=1000mg/day; 2nd increase 1250 mg/day)
Arm/Group | Vatalanib
Serious Adverse Events (participants affected / at risk) | 51/153
Other Adverse Events (participants affected / at risk) | 134/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatalanib (N=153)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8)
Hemoglobin decreased (Blood and lymphatic system disorders) | 43 (48)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 21 (23)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 30 (33)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 28 (31)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 5 (5)
Death NOS (General disorders) | 2 (2)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 35 (41)
Fever (General disorders) | 8 (8)
Hypothermia (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Sudden death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Duodenal infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 10 (11)
Alkaline phosphatase (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 12 (13)
Blood bilirubin increased (Investigations) | 6 (6)
Cardiac troponin I increased (Investigations) | 1 (1)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 7 (8)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
INR increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 26 (30)
Platelet count decreased (Investigations) | 41 (47)
Serum cholesterol increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 11 (12)
Blood glucose increased (Metabolism and nutrition disorders) | 13 (16)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 8 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (9)
Serum calcium decreased (Metabolism and nutrition disorders) | 12 (13)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (6)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (9)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 6 (6)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 14 (14)
Extrapyramidal disorder (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 10 (10)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 10 (12)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (9)
Hypotension (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatalanib (N=153)
Blood disorder (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12)
Hemoglobin decreased (Blood and lymphatic system disorders) | 121 (324)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Transfusion: pRBCs for pediatric BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 4 (4)
Myocardial ischemia (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 4 (6)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (3)
Endocrine disorder (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 23 (28)
Diarrhea (Gastrointestinal disorders) | 45 (71)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 8 (9)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 7 (8)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (8)
Hemorrhoids (Gastrointestinal disorders) | 3 (4)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 80 (135)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 52 (70)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 6 (8)
Death NOS (General disorders) | 2 (2)
Edema limbs (General disorders) | 15 (21)
Fatigue (General disorders) | 116 (233)
Fever (General disorders) | 12 (16)
Gait abnormal (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (1)
Pain (General disorders) | 11 (13)
Visceral edema (General disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2)
Duodenal infection (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 5 (5)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 7 (7)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (6)
Alanine aminotransferase increased (Investigations) | 27 (41)
Alkaline phosphatase increased (Investigations) | 13 (18)
Aspartate aminotransferase increased (Investigations) | 25 (36)
Blood bilirubin increased (Investigations) | 8 (12)
Coagulopathy (Investigations) | 2 (3)
Creatinine increased (Investigations) | 9 (14)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3)
INR increased (Investigations) | 3 (4)
Laboratory test abnormal (Investigations) | 7 (8)
Leukocyte count decreased (Investigations) | 15 (29)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 88 (198)
Pancreatic enzymes decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 100 (226)
Serum cholesterol increased (Investigations) | 4 (7)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 15 (15)
Anorexia (Metabolism and nutrition disorders) | 26 (36)
Blood glucose increased (Metabolism and nutrition disorders) | 37 (70)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Iron overload (Metabolism and nutrition disorders) | 3 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 12 (15)
Serum calcium decreased (Metabolism and nutrition disorders) | 11 (16)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (9)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (9)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 15 (17)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 60 (82)
Dysgeusia (Nervous system disorders) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 19 (22)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (5)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2)
Neurological disorder NOS (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (16)
Speech disorder (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (4)
Vagus nerve disorder (Nervous system disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 3 (3)
Euphoria (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 9 (12)
Cystitis (Renal and urinary disorders) | 2 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (4)
Kidney pain (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 30 (47)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 37 (51)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Rash desquamating (Skin and subcutaneous tissue disorders) | 20 (25)
Skin disorder (Skin and subcutaneous tissue disorders) | 9 (9)
Sweating (Skin and subcutaneous tissue disorders) | 6 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Hematoma (Vascular disorders) | 3 (4)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (15)
Hypotension (Vascular disorders) | 4 (4)
Thrombosis (Vascular disorders) | 2 (3)
Vascular disorder (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less